CLINICAL TRIAL: NCT01569919
Title: A Phase II Trial to Assess the Safety, Immunological Activity of TroVax® Plus Pemetrexed/Cisplatin in Patients With Malignant Pleural Mesothelioma
Brief Title: A Phase II Trial to Assess TroVax® Plus Chemotherapy in Patients With Malignant Pleural Mesothelioma
Acronym: SKOPOS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wales Cancer Trials Unit (Other)
Collaborators: Velindre NHS Trust (Other Government); June Hancock Mesothelioma Research Fund (Unknown); Velindre Cancer Centre Stepping Stones Appeal (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/VCC/0049; 2010-023230-22 (EudraCT Number)
Record Dates: First submitted 2012-03-28; First posted 2012-04-03 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Malignant; Pleural; Mesothelioma
Keywords: Phase II; Single arm; Vaccine
MeSH Terms: conditions — Mesothelioma | interventions — TroVax; Pemetrexed; Cisplatin; Vitamin B 12; Folic Acid; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TroVax® (Experimental): In this single-arm study, all participants will receive 9 injections of the TroVax® vaccine, plus standard cisplatin and pemetrexed chemotherapy.
  Interventions: Biological: TroVax®; Drug: Pemetrexed; Drug: Cisplatin; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid; Drug: Dexamethasone

INTERVENTIONS:
Biological: TroVax® — Dose of 1 x 10^9 TCID 50/ml, in 1ml, given on day 1 of weeks 1, 3, 6, 9, 12, 15, 18, 21, 24.
Drug: Pemetrexed — 500 mg/m^2 over 10 mins, given on day 3 of weeks 4, 7, 10, 13.
Drug: Cisplatin — 75mg/m^2 over 1 hour, given on day 3 of weeks 4, 7, 10, 13
Dietary Supplement: Vitamin B12 — 1000μg intramuscular, Day 2 of weeks 3 and 12
Dietary Supplement: Folic Acid — 400μg oral daily from Day 2 of week 3 to Day 2 of week 16
Drug: Dexamethasone — 4mg BD, Days 2-6 of weeks 4, 7, 10, 13

SUMMARY:
This study is for patients with malignant mesothelioma of the lung lining (called pleura) who are planning to have pemetrexed-cisplatin chemotherapy.

We are investigating whether giving a vaccine called TroVax® with pemetrexed-cisplatin chemotherapy is both safe and potentially beneficial in patients with mesothelioma. This vaccine has been used in combination with chemotherapy in other types of cancer and has been shown to be safe. Cancer vaccines work by stimulating the person's immune system to fight the disease, in a similar way to the immune system fighting infection. In laboratory experiments, the vaccine has been shown to stimulate an immune response to a particular protein widely found on mesothelioma cells called 5T4. In patients with mesothelioma it is hoped that the vaccine will stimulate the immune system to attack mesothelioma cells carrying the 5T4 protein.

Pemetrexed-cisplatin chemotherapy is currently seen as the best treatment for patients with mesothelioma, and this is why we plan to combine it with the vaccine. It is hoped that the combination of the TroVax® vaccine and chemotherapy is more beneficial than chemotherapy alone.

Pemetrexed-cisplatin will be given into a vein in the arm (intravenously) every 3 weeks. The TroVax® vaccine will be given as an injection into the shoulder muscle (intramuscularly) 3 weeks before chemotherapy starts, one week before chemotherapy starts, then every 3 weeks. Each participant will receive 4 chemotherapy and 9 vaccine treatments if they complete the planned trial schedule. We aim to recruit 26 patients into the trial over a two year period. If this study shows that pemetrexed-cisplatin chemotherapy plus the TroVax® vaccine is safe and beneficial in terms of stimulating the immune system, the combination will be tested further in larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent obtained from the patient in accordance with the local regulations
* Locally advanced or metastatic, histologically or cytologically proven MPM
* Aged 18 years or over
* WHO performance status 0-1 (Appendix I)
* Life expectancy > 6months
* Haemoglobin ≥ 12 g/dl, total white cell count ≥ 3 x 10^9/L, neutrophil count > 1.5 x 10^9/L, lymphocyte count ≥1 x 10^9/L, monocyte count <0.8 x 10^9/L platelet count >100 x 10^9/L and <400 x 10^9/L. Blood transfusion is allowed.
* Adequate renal function: Creatinine ≥ 50 mL/min as measured by EDTA or 60mL/min as measured by the Cockcroft-Gault formula
* Adequate liver function: ALT, AST and bilirubin < 2 times the upper limit of normal
* At least four weeks from any previous therapy including surgery, or radiotherapy
* Able to comply with the protocol
* Women must be either post-menopausal, or rendered surgically sterile or, if of child-bearing potential, must have a negative pregnancy test prior to trial entry. Two reliable forms of contraception (oral contraception and a barrier method) must be used by all participants while they are being treated with the TroVax® vaccine. Females must continue to use this level of contraception for 3 months following the last trial treatment, and male patients must continue for 1 month.

Exclusion Criteria:

* Serious infections within the 28 days prior to entry to the trial.
* Prior TroVax® treatment
* Previous chemotherapy for MPM
* Major surgery or radiation therapy completed ≤ 4 weeks prior to enrolment
* Prior radiopharmaceuticals (strontium, samarium) less than 8 weeks prior to enrolment
* Participation in any other clinical trial of a licensed or unlicensed drug within the previous 30 days
* History of prior malignant disease unless patient has been disease-free for at least 3 years or the tumour was a non-melanoma skin cancer or early cervical cancer
* Autoimmune disease including systemic Lupus Erythematosis, Grave's disease, Hashimoto's thyroiditis, multiple sclerosis, insulin dependent diabetes mellitus or systemic (non-joint) manifestations of rheumatoid disease
* Clinical significant cardiac failure or a measured ejection fraction of <40%
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgement of the investigator, would make the patient inappropriate for entry into this study.
* Chronic corticosteroid use unless prescribed as replacement therapy in the case of adrenal insufficiency, or other immunosuppressive agents. Dexamethasone is allowed as part of trial treatment.
* Cerebral metastases
* History of allergic response to previous vaccine vaccinations
* Known allergy to egg proteins
* Known to test positive for HIV or hepatitis B or C
* Pregnancy or lactation
* Prior history of organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Immune response to 5T4 and MVA antigens as measured by intracellular cytokine staining (ICCS) | 34 weeks
  To evaluate whether TroVax® is active in the treatment of MPM. This will be assessed by measuring the cellular or humoral anti-5T4 immune responses following treatment with TroVax® given in combination with Pem/Cis.

SECONDARY OUTCOMES:
Safety and tolerability | 34 weeks
  To investigate the safety and tolerability of TroVax® in combination with Pem/Cis. This will be assessed from toxicity data, SAE reports and dose of chemotherapy received
Clinical activity in terms of PFS, ORR and OS | 1 year
  To assess secondary measures of clinical activity, including progression-free survival (PFS), objective response rate (ORR), overall survival (OS) at 6 months and 1 year
Relationship between immune response and clinical response | 1 year
  To explore the relationship between immune response (antibody and cellular responses against the tumour 5T4 and the MVA viral vector) and clinical response (PFS, ORR, OS).
Identify potential predictors of treatment benefit | 1 year
  To investigate the utility of (a) baseline platelet levels, (b) baseline monocyte levels and (c) baseline haemoglobin as predictors of treatment benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Jason F Lester, FRCR, MRCP, Principal Investigator — Velindre Cancer Centre
Locations (1):
- Velindre Cancer Centre, Cardiff, South Wales, United Kingdom